CLINICAL TRIAL: NCT06033352
Title: Comparison of the Efficacy of Potassium-titanyl Phosphate (KTP) Laser vs KTP Laser Combined With Ivermectin 1% Cream for Facial Rosacea: a Randomized Split-face Trial
Brief Title: Potassium-titanyl Phosphate (KTP) Laser vs KTP Laser and Ivermectin Cream for Facial Rosacea
Acronym: KIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-D0015
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Rosacea
Keywords: Rosacea; Laser; Ivermectin
MeSH Terms: conditions — Rosacea | interventions — Lasers, Solid-State; Ivermectin

STUDY DESIGN:
Intervention Model Description: 1:1 within-patient (split-face) random allocation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser and cream (Experimental)
  Interventions: Device: KTP laser; Drug: Ivermectin 1% cream
- Laser alone (Active Comparator)
  Interventions: Device: KTP laser

INTERVENTIONS:
Device: KTP laser — Treatment with KTP 532 nm laser. Laser fluence depends on erythema intensity and ranges from 7.0 J/cm2 to 11 J/cm2 with a 4-11 mm spot size and 8-12 ms pulse duration.
Drug: Ivermectin 1% cream — Application of ivermectin 1% cream 1x/day. Interruption for 4 days in case of irritation/redness.
  Arms: Laser and cream

SUMMARY:
Rosacea is a frequent chronic inflammatory disease affecting mainly the face but also eyes and scalp. Rosacea is classified into 3 types: erythemato-teleangiectatica, papulopustulosa and phymatosa. Treatments depend on the type and include topical and systemic antibiotics, azelaic acid, topical ivermectin, topical brimonidine, systemic isotretinoin as well as intense pulsed light (IPL) and laser therapies.

For treatment of telangiectasia and redness, laser and IPL therapies are the first choice. Vascular lasers, such as pulsed dye lasers (PDL) and potassium-titanyl phosphate (KTP) lasers as well as IPL, have demonstrated good efficacy in reduction of erythema and telangiectasias in patients with rosacea. However, these treatments are expensive and mostly not covered by the health insurance. Therefore, for patients it is important to receive the maximal effect and improvement after each single laser session.

Ivermectin is a semi-synthetic derivative of avermectin and has an anti-inflammatory effect as well as an antiparasitic effect on demodex mite. The latter is playing an important pathogenetic role in rosacea.

This randomized controlled study aims to compare the effect of KTP laser in combination with ivermectin 1% cream vs KTP laser alone in patients with facial rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin type I-IV
* Presence of facial erythematous rosacea or mild papulopustular rosacea with permanent erythema
* Informed consent signed

Exclusion Criteria:

* History of adverse events related to KTP laser therapy
* Pregnant or breastfeeding women
* Intention to become pregnant during the course of the study
* History of intolerance or allergic reaction to ivermectin 1% cream or one of the ingredients
* Ongoing treatment for skin cancer
* Ongoing treatment with strong inhibitors of P-glycoprotein (P-gp) and CYP3A4 (e.g., itraconazole, voriconazole, posaconazole, clarithromycin, cobicistat)
* Ongoing treatment with substances with a narrow therapeutic range whose excretion depends substantially on P-gp (e.g. digoxin, ciclosporin)
* Inability to understand the study content

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of laser and cream vs laser alone in reducing erythema as assessed by NEI | 16 weeks
  Any relative decrease of erythema on the side treated with KTP laser and ivermectin 1% cream vs laser alone as assessed by Normalized Erythema Index (NEI), ranging from 0 to 80, with higher values indicating a worst erythema.

SECONDARY OUTCOMES:
Efficacy of laser and cream vs laser alone in reducing erythema as assessed by SRI | 16 weeks
  Any relative decrease of erythema on the side treated with KTP laser and ivermectin 1% cream vs laser alone as assessed by Skin Redness Index (SRI), ranging from 1 to 4, with higher score indicating a worst erythema.
Efficacy of laser and cream vs laser alone in reducing erythema as assessed by CEA | 4, 8, 12, 16 weeks
  Any decrease of erythema on the side treated with KTP laser and ivermectin 1% cream vs laser alone as assessed by Clinical Erythema Assessment (CEA), ranging from 0 to 4, with higher score indicating a worst erythema.
Efficacy of laser and cream vs laser alone in the clinical improvement of skin lesions as assessed by PGA | 4, 8, 12, 16 weeks
  Any change of skin lesions on the side treated with KTP laser and ivermectin 1% cream vs laser alone as assessed by 6-point Physician Global Assessment (PGA), ranging from 0 to 5, with higher score indicating a better outcome.
Patient's satisfaction related to laser and cream vs laser alone in the improvement of skin lesions as assessed by VAS | 4, 8, 12, 16 weeks
  Any difference of patient's satisfaction for the improvement of skin lesions on the side treated with KTP laser and ivermectin 1% cream vs laser alone as assessed by a 9-point anchored visual analogue scale (VAS), ranging from -4 to +4, with negative scores indicating a worsening of condition, with 0 indicating no difference and with positive scores indicating an improvement.
Efficacy of laser and cream vs laser alone in reducing telangiectasia severity as assessed by TGS | 4, 8, 12, 16 weeks
  Any change of telangiectasia severity on the side treated with KTP laser and ivermectin 1% cream vs laser alone as assessed by telangiectasia grading scale (TGS), ranging from 0 to 3, with higher score indicating a worst telangiectasia severity.
Efficacy of laser and cream vs laser alone in reducing papules and papulopustules | 4, 8, 12, 16 weeks
  Any change in the number of papules and papulopustules on the side treated with KTP laser and ivermectin 1% cream vs laser alone.
Efficacy of laser and cream vs laser alone in reducing face swelling as assessed by the patient | 4, 8, 12, 16 weeks
  Any change in the number of days of face swelling on the side treated with KTP laser and ivermectin 1% cream vs laser alone, as assessed by the patient
Efficacy of laser and cream vs laser alone in reducing face redness as assessed by the patient | 4, 8, 12, 16 weeks
  Any change in the number of days of face redness on the side treated with KTP laser and ivermectin 1% cream vs laser alone, as assessed by the patient.
Efficacy of laser and cream vs laser alone in reducing face purpura as assessed by the patient | 4, 8, 12, 16 weeks
  Any change in the number of days of face purpura on the side treated with KTP laser and ivermectin 1% cream vs laser alone, as assessed by the patient.

OTHER OUTCOMES:
Incidence of observed side-effects | 16 weeks
  Cumulative number of observed treatment side-effects.
Incidence of observed adverse events | 16 weeks
  Cumulative number of observed treatment adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Heidemeyer, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Department of dermatology, University Hospital Inselspital, Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No